CLINICAL TRIAL: NCT03268226
Title: Open Label, Prospective, Exploratory Study to Investigate the Effect of Inhaled CHF5993 pMDI on Central and Peripheral Airway Dimensions in COPD Patients by Functional Respiratory Imaging
Brief Title: Functional Respiratory Imaging Study (FRI)
Acronym: FRI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCD-05993AA1-16; 2017-000438-79 (EudraCT Number)
Record Dates: First submitted 2017-08-23; First posted 2017-08-31 (Actual); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Beclomethasone

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CHF5993 (Experimental): Beclometasone dipropionate/Formoterol Fumarate/Glycopyrronium Bromide administered via pMDI
  Interventions: Drug: Beclometasone dipropionate/Formoterol Fumarate/Glycopyrronium

INTERVENTIONS:
Drug: Beclometasone dipropionate/Formoterol Fumarate/Glycopyrronium — An inhaled dose of CHF 5993 pMDI 100+6+12.5 μg twice a day (Total daily dose: BDP 400 μg / FF 24 μg / GB 50 μg)

SUMMARY:
The purpose of this study is to evaluate the effect of inhaled extrafine CHF5993 pMDI on airway volumes, and resistance, by Functional Respiratory Imaging (FRI), in COPD patients

ELIGIBILITY:
Inclusion Criteria:

1. Subject's written informed consent obtained prior to any study-related procedure.
2. Male or Female COPD patients aged ≥ 40 years.
3. Smoking history: of at least 10 pack-years (pack-year= number of cigarettes per day x number of years/20).
4. Smoking status: current or ex-smokers. Previous smokers are defined as those who have stopped smoking for at least 24 weeks prior to screening visit. (Pipe and/or cigar and/or e-cigarettes smoking cannot be used to calculate pack-year history). If the subjects undergo smoking cessation therapy, it must be completed 3 months prior to study entry.
5. Patients with documented COPD at least 12 months according to GOLD 2017.
6. Post-bronchodilator (BD) decreased Tiffeneau index: FEV1/FVC < 0.70.
7. Patients who present post- BD FEV1 less than 50 % of predicted.
8. Patients who present (Functional residual capacity) FRC ≥120% predicted.
9. Patients who present CAT assessment ≥10.
10. Patients on stable respiratory medications for at least 3 months prior to screening with non extrafine extemporary triple combination. The possible combination therapies prior to screening are:

    * fluticasone plus salmeterol plus tiotropium
    * fluticasone plus salmeterol plus glycopyrronium
    * fluticasone plus salmeterol plus umeclidinium
    * fluticasone plus vilanterol plus tiotropium
    * fluticasone plus vilanterol plus glycopyrronium
    * fluticasone plus vilanterol plus umeclidinium;
11. Body Mass Index (BMI) between 18.0 and 32.0 kg/m2 (extremes included) at the screening visit..
12. Ability to understand the study procedures and the risks involved and ability to be trained with pMDI training inhalers to use the devices correctly.
13. WOCBP fulfilling one of the following criteria:

    1. WOCBP with fertile male partners: they and/or their partner must be willing to use a highly effective birth control method from the signature of the informed consent and until the follow-up visit or
    2. WOCBP with non-fertile male partners (contraception is not required in this case).

    For the definition of WOCBP and of fertile men and the list of highly effective birth control methods, refer the CTFG guidance for more detailed information
14. Female patients of non-childbearing potential defined as physiologically incapable of becoming pregnant (i.e. post-menopausal or permanently sterile; e.g. amenorrehic for ≥12 consecutive months without alternative medical cause). Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy (40). If indicated, as per investigator's request, post-menopausal status may be confirmed by follicle-stimulating hormone levels (according to local laboratory ranges).

Exclusion Criteria:

1. Pregnant or lactating women.
2. Patients with history or current diagnosis of asthma.
3. Medical history or current diagnosis of allergic rhinitis or atopy (atopy which may have risen contra-indications or impacted the efficacy of the study treatment according to Investigator's judgment).
4. Patients requiring use of the following medications:

   1. Systemic steroids for COPD exacerbation in the 4 weeks prior to screening;
   2. Patients with a moderate or severe COPD exacerbation [i.e. resulting in the use of systemic corticosteroids (oral/IV/IM) and/or or antibiotics or need for hospitalisation within 6 weeks prior to screening];
   3. A course of antibiotics for COPD exacerbation longer than 7 days in the 4 weeks prior to screening;
   4. c-Phosphodiesterase-4 (PDE-4) inhibitors in the 4 weeks prior to screening;
   5. Use of antibiotics for a lower respiratory tract infection (e.g. pneumonia) in the 4 weeks prior to screening;
5. Patients treated with non-cardio-selective β-blockers in the week prior to screening.
6. Patients treated with long-acting anti-histamines unless taken at stable regimen at least 2 months prior to screening and to be maintained constant during the study.
7. Patients requiring long term (at least 12 hours daily) oxygen therapy for chronic hypoxemia.
8. Known respiratory disorders other than COPD which may impact the efficacy of the study treatment according the Investigator's judgment. (This could include but is not limited to α-1 antitrypsin deficiency, active tuberculosis, bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension and interstitial lung disease).
9. Lung cancer or history of lung cancer: patients with a diagnosis of lung cancer or a history of lung cancer.
10. Lung resection: subjects with a history of lung volume resection.
11. Subjects who have a cardiovascular condition such as, but not limited to unstable ischemic heart disease, NYHA Class III/IV left ventricular failure, acute ischemic heart disease in the last year prior to study screening, which may impact the safety of the subject or the evaluation of the result of the study according to the Investigator's judgment; history of atrial fibrillation, history of sustained and non sustained cardiac arrhythmias diagnosed within 24 weeks prior to study entry not controlled with therapy.
12. ECG criteria: any clinically significant abnormal 12-lead ECG that in the Investigator's opinion would affect the efficacy or safety evaluation or place the patients at risk. Male patients with a QTcF >450ms and female patients with a QTcF >470ms at screening and/or baseline visits are not eligible.
13. Medical history or current diagnosis of narrow-angle glaucoma, clinically relevant prostatic hypertrophy or bladder neck obstruction that in the opinion of the Investigator would have prevented use of anticholinergic agents.
14. History of hypersensitivity to M3 antagonists, β2-agonist, corticosteroids or any of the excipients contained in any of the formulations used in the study which may raise contra-indications or impacted the efficacy of the study treatment according to the Investigator's judgment.
15. Clinically significant laboratory abnormalities indicating a significant or unstable concomitant disease which may have impacted the efficacy or the safety of the study treatment according to Investigator's judgment.
16. Patients with serum potassium levels < 3.5 mEq/L (or 3.5 mmol/L).
17. Unstable concurrent disease: e.g. uncontrolled hyperthyroidism, uncontrolled diabetes mellitus or other endocrine disease; uncontrolled gastrointestinal disease (e.g. active peptic ulcer); uncontrolled neurological disease; uncontrolled hematological disease; uncontrolled autoimmune disorders, or other which may impact the feasibility of the results of the study according to Investigator's judgment.
18. History of alcohol abuse and/or substance/drug abuse within 12 months prior to screening.
19. Drugs with hepatoxic potential: Patients receiving treatment with any drug known to have a well defined potential for hepatotoxicity (e.g. isoniazide, nimesulide, ketoconazole) within the previous 3 months before the screening visit.
20. Changes in dose, schedule, formulation or product of oral xanthine derivatives (e.g. Theophylline) in the month prior screening visit.
21. Participation in an investigational trial: patients who have received any investigational drug within the 30 days (60 days for biologics) before the screening visit or a more appropriate time as determined by the investigator (e.g. approximately 5 half-lives of the investigational drug whatever is longer).
22. Treatment with strong CYP3A inhibitors (e.g. erythromycin, itraconazole) within 4 weeks prior to study entry.
23. Serology at the screening positive for HIV1 or HIV2 and positive results for Hepatitis which indicates acute or chronic Hepatitis B (i.e. positive HB surface antigen HBsAg, positive and/or positive HB core antibody anti-HBc) or Hepatitis C (positive HCV antibody).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Specific image-based airway volumes (siVaw) | Change from baseline at 24 Weeks.
  CT-based airway volumes normalized by the lung volume
Specific image-based airway resistance (siRaw) | Change from baseline at 24 Weeks.
  CFD-based airway resistance normalized by the lung volume

SECONDARY OUTCOMES:
Internal Airflow Distribution | On Week 0, Week 12, and on Week 24
  calculated using thorax HRCT
Air Trapping | On Week 0, Week 12, and on Week 24
  calculated using thorax HRCT
Emphysema | On Week 0, Week 12, and on Week 24
  calculated using thorax HRCT
Airway Wall Volume | On Week 0, Week 12, and on Week 24
  calculated using thorax HRCT
Blood vessel density | On Week 0, Week 12, and on Week 24
  calculated using thorax HRCT
Ventilation/perfusion matching | On Week 0, Week 12, and on Week 24
  calculated using thorax HRCT
Aerosol Deposition | On Week 0, Week 12, and on Week 24
  calculated using thorax HRCT
Functional Dyspnea | On Week 0, Week 12, and on Week 24
  mMRC dyspnea scale
Quality of life | On Week 0, Week 12, and on Week 24
  Saint George Respiratory Questionnaire (SGRQ)
CAT score | On Week 0, Week 12, and on Week 24
  8-items unidimensional questionnaire
Dyspnea | On Week 0, Week 12, and on Week 24
  Borg CR10
Dynamic lung volumes | On Week 0, Week 12, and on Week 24
  calculated using spirometry
Static lung volumes | On Week 0, Week 12, and on Week 24
  calculated using body plethysmography
airway resistances | On Week 0, Week 12, and on Week 24
  calculated using body plethysmography

OTHER OUTCOMES:
exercise tolerance | On Week 0, Week 12, and on Week 24
  cycling endurance test (CET)

CONTACTS AND LOCATIONS:
Locations (5):
- Belgium (4):
  - SGS CPU Antwerpen, Antwerp
  - AZ Saint-Maarten, Duffel
  - Centre medical Erpent - Residence, Erpent
  - Heilige Familie AZ, Reet
- National Koranyi Institute for TB and Pulmonology, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Study Record on EU Clinical Trials Register including results. — https://www.clinicaltrialsregister.eu/ctr-search/trial/2017-000438-79/results